CLINICAL TRIAL: NCT03950063
Title: Cutibacterium Acnes in Bone and Joint Infections
Acronym: CaBJI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA18027
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Prosthesis and Bone Infections; Cutibacterium Acnes
Keywords: Cutibacterium acnes Prosthesis; Bone Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cutibacterium acnes bone infections: Patients with Cutibacterium acnes orthopedic material infections

SUMMARY:
Prosthetic Joint Infections (PJIs) are increasing with the use of orthopedic devices on an ageing population. Cutibacterium acnes is a commensal organism that plays an important role in the ecosystem healthy human skin, yet this species is also recognized as a pathogen in foreign body infection: endocarditis, prostatitis and specifically in PJIs. C. acnes is able to escape the immune system. This phenomenon could reflect two bacterial behavior: the bacterial internalization by host cells and the biofilm formation.

DETAILED DESCRIPTION:
The aim of the study is to evaluate specific pathogenicity factors (ability to internalize bone cells and ability to form a biofilm) of bacteria derived from clinical strains of C. acnes isolated from bone infections on orthopedic material.

ELIGIBILITY:
Inclusion Criteria:

* bone infection with C. acnes,
* isolation of the strain,
* presence of a single species,
* conservation of a viable strain,
* patients over 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cutibacterium acnes bone infections
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Internalization capacity of C. acnes strains | Day 0
  C. acnes strains will be cultured for 5 days in rich medium at 37°C in anaerobic conditions. Then, the bacteria will be co cultured with bone cells (osteoblast) and bacteria will be internalized by the bone cells. After killing bacteria stayed outside of the cells with an antibiotic and lysis of the cells, the number of bacteria internalized will be counted on agar plate.
Biofilm capacity of C. acnes strains | Day 0
  C. acnes strains will be cultured for 5 days in rich medium at 37°C in anaerobic conditions. Then, the biofilm biomass will be evaluated by Crystal violet staining. The amount of biofilm will be evaluated by absorbance (optic density by spectrophotometry).

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France